CLINICAL TRIAL: NCT05249361
Title: Correlation Between Functional Capacity and Functional Capability in Patients With Duchenne Muscular Dystrophy-A Longitudinal Study
Brief Title: Correlation Between Functional Capacity and Functional Capability in Duchenne Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Other Study IDs: 2022-05-136
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Accelerometer; ActiGraph; DEXA; muscle ultrasound
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duchenne Muscular Dystrophy: Children aged 5 to 18 years with Duchenne muscular dystrophy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study investigates the correlation between assessments measuring functional capacity and functional capability in patients with Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
This study is a prospective single-arm observational study, with a total of two visits for one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 to 18 years diagnosed with Duchenne muscular dystrophy through genetic testing
2. Children who understand the contents of this research and can properly conduct the research

Exclusion Criteria:

1. Requiring daytime ventilator assistance or using invasive mechanical ventilation through tracheostomy (Non-invasive mechanical ventilation such as positive pressure ventilation at night is allowed)
2. History of peripheral nerve damage
3. History of major surgery within 12 weeks or if major surgery is expected during the test period
4. History of central nervous system disorders (eg, cerebral infarction, spinal cord injury)
5. Having difficulties in conducting this study due to cognitive decline.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Asian patients of Duchenne muscular dystrophy, who live in South Korea and visited the Samsung medical center in Gangnam-gu, Seoul.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between physical activity(VM) and muscle quantitative index | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in muscle quantitative measures of upper and lower extremities from baseline to 48-week. The activity counts will be measured with ActiGraph wgt3x-bt worn on patient's dominant ankle and wrist. Accelerometers recorded acceleration in three orthogonal axes (x, y, z) at 30 Hz. Accelerometer recordings were uploaded to ActiLife software, integrated into 15-second epochs, and converted into an omnidirectional acceleration estimate, or vector magnitude (VM), calculated as the square root of the sum of the triaxial signals squared.
  The muscle quantitative will be measured with Microfet2. Muscle quantitative of upper extremity is the sum of the flexion and extension of both elbows and lower extremity is the sum of both knee flexion and extension and bilateral ankle dorsiflexion.

SECONDARY OUTCOMES:
Correlation between physical activity and Vignos scale | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in Vignos scale score from baseline to 48-week. On the Vignos scale, the grade ranges from 1 to 10; 1 means that the patient is able to walk and climb stairs without assistance, while 10 means that the patient is bed-bound
Correlation between physical activity and Brooke scale | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in Brooke scale score from baseline to 48-week. The grades on the Brooke scale range from 1 to 6; 1 means that the patient is able to start with arms at the sides and can abduct the arms in a full circle until they touch above the head, while 6 means that they are unable to raise their hands to their mouth and have no useful function of the hands.
Correlation between physical activity and 6MWT(6-minute walking test) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in 6MWT results from baseline to 48-week. The 6MWT assesses distance walked over 6 minutes.
Correlation between physical activity and NSAA(The North Star Ambulatory Assessment) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in NSAA scores from baseline to 48-week. The NSAA is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD). It includes several items assessing abilities that are necessary to remain functionally ambulant, items assessing abilities, such as head raise and standing on heels that can be partly present in the early stages of the disease and a number of activities such as hopping.
  Each item can be scored on a 3 point scale using simple criteria: 2 -Normal achieves goal without any assistance; 1 -Modified method but achieves goal independent of physical assistance from another person; 0 -Unable to achieve independently.
  A total score can be achieved by summing the scores for all the individual items. The score can range from 0, if all the activities are failed, to 34, if all the activities are achieved.
Correlation between physical activity and PUL(Performance of Upper Limb module for DMD) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in PUL scores from baseline to 48-week.
  The PUL includes 22 items with an entry item to define the starting functional level (which corresponds to the Brooke scale) and 21 items subdivided into shoulder level (4 items), elbow level (9 items), and distal (i.e., wrist and fingers) level (8 items). For weaker patients, a low score on the entry item (i.e., less than 4 point of Item A) means that shoulder-level items do not need to be performed. Each dimension can be scored separately with a maximum score of 16 for the shoulder level, 34 for the elbow level, and 24 for the distal level. A total score can be achieved by adding the three-level scores, with a maximum global score of 74 points.
Correlation between physical activity and PEDI-CAT(the Pediatric Evaluation of Disability Inventory-Computer Adaptive Test) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in mobility and self-care domain scores of PEDI-CAT from baseline to 48-week.
  Te PEDI-CAT incorporates a computer-adaptive platform with 276 items based on parental or caregiver reporting, and has four domains that cover daily activities, mobility, social/cognitive function, and responsibility. The PEDI-CAT yields a single score scaled from 0 to 100 for both Mobility and Self-care, with higher scores indicating greater function.
Correlation between physical activity and EQ-5D(EuroQol-5D) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in EQ-5D from baseline to 48-week.
  EuroQol EQ-5D is a preference-based HRQOL measurement tool for the five dimensions of 'exercise ability', 'self-management', 'daily activity', 'pain/discomfort', and 'anxiety/depression' in terms of 'no problem', 'somewhat Evaluated on three levels of 'having a problem' and 'having a serious problem', and the overall level was evaluated on a thermometer-shaped 20 cm vertical visual analogue scale with 0 points for the lowest health and 100 points for the highest health status.
Correlation between physical activity and CHQ-PF50(Child Health Questionnaire - Parent form 50 ) | Baseline up to Week 48
  We analyze the correlation between the change in activity counts from baseline to 48-week and the change in EQ-5D from baseline to 48-week.
  The Child Health Questionnaire - Parent form 50 (CHQ-PF50) consists of 50 questions and 12 scales (Physical function, Role/social limitations-physical, Role/social limitations-emotional/ behavioral, Mental health, Self-esteem, Behavior, Bodily pain/discomfort, General health perceptions, Family activities, Parent impact on time, Parent emotional impact) and 2 global items (Global behavior and global general health), 2 summary scores (Physical and a psychosocial summary scores) is a tool to evaluate the quality of life of children. The raw score is converted into a converted score between 0-100, and the higher the score, the better the quality of life.
Correlation between physical activity and quantitative muscle ultrasonography | Baseline up to Week 48
  We analyze the correlation between change in activity from baseline to 48-week and the change in quantitative muscle ultrasonography from baseline to 48-week. We will measure the echogenicity of the muscles at 12 sites including deltoid, biceps brachii, wrist/finger flexors, rectus femoris, tibialis anterior, medial gastrocnemius, masseter, sternocleidomastoid, geniohyoid and diaphragm. The average gray scale of above muscles will be analyzed with ImageJ software (https://imagej.nih.gov).
Correlation between physical activity and DMD upper limb PROM | Baseline up to Week 48
  We analyze the correlation between change in activity from baseline to 48-week and the change in DMD upper limb PROM from baseline to 48-week. DMD upper limb PROM is a patient reported outcome measure designed to assess upper extremity performance in daily life. It includes 32 items and each item will be scored on a 3 point scale: 2-can do task easily; 1-can do tast with difficulty; 0-impossible without help. A total score is the summation of the scores for all individual items. The score can range from 0 to 64.
Correlation between physical activity and Pulmonary function test | Baseline up to Week 48
  We analyze the correlation between change in activity from baseline to 48-week and the change in pulmonary function test from baseline to 48-week. Maximal inspiratory pressure and maximal expiratory pressure will be measured with spirometry (Spirovis, Cosmed Srl, Rome, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-yi Kwon, MD,Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Im YJ, Choe Y, Lee J, Lee J, Do JG, Kwon JY. Quantitative Muscle Ultrasound: A Non-Invasive Biomarker for Monitoring Duchenne Muscular Dystrophy. Muscle Nerve. 2025 Oct;72(4):606-615. doi: 10.1002/mus.28469. Epub 2025 Jul 16. PMID 40671379